CLINICAL TRIAL: NCT03151616
Title: Association of Anticholinergic Risk Scale and Healthcare Resource Use After Elective Noncardiac Surgery: a Population-based Cohort Study
Brief Title: Anticholinergic Risk Scale and Resource Use After Elective Noncardiac Surgery
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dan McIsaac, Associate Scientist, Ottawa Hospital Research Institute
Other Study IDs: DM6
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-10

CONDITIONS: Length of Stay; Anti Cholinergics; Surgical Procedure, Operative; Aged; Epidemiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No anticholinergic exposure: People with an anticholinergic risk scale score of 0
- Moderate anticholinergic exposure: People with an anticholinergic risk scale score of 1-2
  Interventions: Other: anticholinergic risk scale
- High anticholinergic exposure: People with an anticholinergic risk scale score of >=3
  Interventions: Other: anticholinergic risk scale

INTERVENTIONS:
Other: anticholinergic risk scale — Risk summation scale for grading and studying anticholinergic medication exposure
  Groups: High anticholinergic exposure; Moderate anticholinergic exposure

SUMMARY:
This study investigates the association of preoperative anticholinergic medication exposure with healthcare resource utilization in a population-based sample of older patients enrolled in a universal pharmacare program

DETAILED DESCRIPTION:
Multilevel multivariable regression analysis will be used to investigate the adjusted association between preoperative Anticholinergic Risk Scale and postoperative healthcare resource utilization. Sensitivity analyses will be used to evaluate the robustness of the primary analysis.

ELIGIBILITY:
Inclusion Criteria:

* at least 66 years old on the day of surgery
* Intermediate to high risk elective noncardiac surgery

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Population-based sample of people having their first eligible surgery during the study period
Sampling Method: Non-Probability Sample
Enrollment: 244976 (Actual)
Dates: Start 2003-04-01 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2014-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Anticholinergic Exposure | Moderate Anticholinergic Exposure | High Anticholinergic Exposure
Started | 173522 | 38127 | 33327
Completed | 173522 | 38127 | 33327
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Anticholinergic Exposure | Moderate Anticholinergic Exposure | High Anticholinergic Exposure | Total
Number analyzed (Participants) | 173522 | 38127 | 33327 | 244976
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (6) | 74 (6) | 75 (6) | 74 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86587 | 23257 | 20063 | 129907
  Male | 86935 | 14870 | 13264 | 115069

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Number of days in hospital after surgery
Time Frame: date of surgery to date of hospital discharge, or 365 days after surgery, whichever comes first
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | No Anticholinergic Exposure | Moderate Anticholinergic Exposure | High Anticholinergic Exposure
Number analyzed (Participants) | 173522 | 38127 | 33327
Days | 6.8 (9.7) | 7.8 (11.4) | 7.5 (11.3)

2. Secondary Outcome: Costs of Care
Description: Costs related to medical care paid for by the provincial health insurance system
Time Frame: date of surgery up to 90 days after surgery
Measure: Mean (Standard Deviation); unit: Canadian Dollars
Arm/Group | No Anticholinergic Exposure | Moderate Anticholinergic Exposure | High Anticholinergic Exposure
Number analyzed (Participants) | 173522 | 38127 | 33327
Canadian Dollars | 21528 (21645) | 24108 (23342) | 24610 (24679)

3. Secondary Outcome: Institutional Discharge
Description: A discharge location at the end of the surgical episode of care that is not back to the patient's original residence (specifically respite or long term care)
Time Frame: date of surgery to date of hospital discharge, or 365 days after surgery, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | No Anticholinergic Exposure | Moderate Anticholinergic Exposure | High Anticholinergic Exposure
Number analyzed (Participants) | 173522 | 38127 | 33327
Participants | 34724 | 8885 | 7371

4. Secondary Outcome: Mortality
Description: death from any cause
Time Frame: from day of surgery up to 90 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | No Anticholinergic Exposure | Moderate Anticholinergic Exposure | High Anticholinergic Exposure
Number analyzed (Participants) | 173522 | 38127 | 33327
Participants | 3515 | 1154 | 939

5. Secondary Outcome: Hospital Readmission
Description: Acute hospital readmission after discharge from index hospitalization
Time Frame: From the date of hospital discharge to 30 days after the date of discharge
Measure: Count of Participants; unit: Participants
Arm/Group | No Anticholinergic Exposure | Moderate Anticholinergic Exposure | High Anticholinergic Exposure
Number analyzed (Participants) | 173522 | 38127 | 33327
Participants | 10905 | 2981 | 2666

ADVERSE EVENTS:
Time Frame: 1 year
Description: The occurrence of death due to any cause was collected.
  No other adverse events were collected.
Arm/Group | No Anticholinergic Exposure | Moderate Anticholinergic Exposure | High Anticholinergic Exposure
All-Cause Mortality (participants affected / at risk) | 3515/173522 | 1154/38127 | 939/33327
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The data used were not initially collected for research purposes and could be subject to misclassification bias. Our findings are at risk of unmeasured confounding. Administrative data do not accurately capture delirium, so we were unable to provide estimates of the association of the ARS with delirium rates. We chose to use the ARS as our measure of anticholinergic exposure; however, several anticholinergic scales have been described and effect sizes vary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No